CLINICAL TRIAL: NCT02186080
Title: Evaluation of the Effect of Gemigliptin on Metabolic Endotoxemia and Lipemia Induced by High Fat Diet in Patients With Type 2 Diabetes
Brief Title: Effect of Gemigliptin on Metabolic Endotoxemia and Lipemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-1401-089-550
Record Dates: First submitted 2014-07-04; First posted 2014-07-10 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2014-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes mellitus; metabolic endotoxemia; gemigliptin; DPP-4 inhibitor
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — LC15-0444

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemigliptin (Experimental): Gemigliptin 50mg qd added to subjects current diabetes treatment
  Interventions: Drug: Gemigliptin
- Placebo (Placebo Comparator): Placebo (identical in appearance to gemigliptin)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gemigliptin
  Other Names: Zemiglo
  Arms: Gemigliptin
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is an exploratory study on the metabolic endotoxemia associated with type 2 diabetes. The investigators will measure systemic endotoxin level and lipid level after ingestion of high fat diet to evaluate the effect of gemigliptin, a DPP-4 inhibitor, on metabolic endotoxemia and lipemia induced by high fat diet.

DETAILED DESCRIPTION:
Study subjects will be allocated to either gemigliptin or placebo. After 4 weeks of treatment and 2 weeks of wash out period, all subjects will be switched to the opposite arm.

The subjects will be tested oral fat tolerance test and adipose tissue needle biopsy(only for the subjects who agreed to participate donate adipose tissue) at 3 time points: the start of 1st treatment, end of 1st treatment and end of 2nd treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age from 20 to 75
* At least 6 months from the diagnosis of type 2 diabetes
* Current diabetes treatment: life style modification and/or metformin and/or sulfornylurea
* No change of the diabetes treatment (drug number and dossage) in recent 3 months
* HbA1c 6.5% to 10%

Exclusion Criteria:

* Recent cardiovascular event in 6 months
* Concurrent use of statin or fibrate or ezetimibe
* Renal failure, chronic liver disease
* Pregnancy or lactation
* Use of other DPP-4 inhibitor or GLP-1 analogue in recent 3 months

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Difference between baseline and peak serum LPS | serum LPS before high fat diet and 15 min, 30 min, 1 hr, 2 hr, 3 hr, 4 hr after high fat diet
  The increment of serum LPS after ingestion of high fat diet

SECONDARY OUTCOMES:
Fasting serum LPS level | After 10 hrs of fasting
  Compare fasting LPS level between treatment group
Incremental AUC of serum LPS during oral fat tolerance test | serum LPS before high fat diet and 15 min, 30 min, 1 hr, 2 hr, 3 hr, 4 hr after high fat diet
  Calculated incremental AUC of serum LPS
Difference between baseline and peak serum triglyceride level | serum TG before high fat diet and 15 min, 30 min, 1 hr, 2 hr, 3 hr, 4 hr after high fat diet
  The increment of serum TG after ingestion of high fat diet
Incremental AUC of serum triglyceride level during oral fat tolerance test | serum TG before high fat diet and 15 min, 30 min, 1 hr, 2 hr, 3 hr, 4 hr after high fat diet
  Calculated incremental AUC of serum TG
Difference between baseline and peak serum apolipoprotein-B48 | serum apolipoprotein-B48 before high fat diet and 15 min, 30 min, 1 hr, 2 hr, 3 hr, 4 hr after high fat diet
  The increment of serum apolipoprotein-B48 after ingestion of high fat diet
Incremental AUC of serum apolipoprotein-B48 during oral fat tolerance test | serum apolipoprotein-B48 before high fat diet and 15 min, 30 min, 1 hr, 2 hr, 3 hr, 4 hr after high fat diet
  Calculated incremental AUC of serum apolipoprotein-B48
Serum level of inflammatory markers (CRP, TNF-alpha, IL-6) | After 10 hr of fasting
  Compare serum level of inflammatory markers between treatment groups
mRNA expression level of inflammatory markers in the adipose tissue | After high fat diet ingestion
  Compare mRNA expression level of inflammatory markers

CONTACTS AND LOCATIONS:
Overall Officials: Young Min Cho, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No